CLINICAL TRIAL: NCT00243789
Title: A Double-Blinded Randomized Placebo Controlled Study of Daily Pentoxifylline as a Rescue Treatment in DMD
Brief Title: Study of Daily Pentoxifylline as a Rescue Treatment in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Study Chair, CINRG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNMC0705
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne; Genetic; Muscular Dystrophy; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pentoxifylline
  Interventions: Drug: Pentoxifylline
- 2 (No Intervention): Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Participants will be randomized to receive either pentoxifylline or placebo in addition to their stable steroid therapy. Active drug and placebo preparations will be supplied as gel capsules of identical size, appearance and taste. Active drug capsules will contain one 400 mg time-release pentoxifylline tablet and inert filler. Placebo capsules will contain inert filler.
  Based on weight at screening, <30 mg will receive 1 400 capsule/day; 30-49 kg will receive two 400 capsules/day; 50 kg or greater will receive three 400 mg capsules/day.
  Other Names: Trental
  Arms: 1

SUMMARY:
The purpose of this study is to see if male children with Duchenne muscular dystrophy (DMD) have changes in strength when given the drug Pentoxifylline as a rescue treatment. A total of 64 subjects are expected to participate through all other centers of the Cooperative International Neuromuscular Research Group (CINRG) worldwide.

The primary purpose of this study is to see whether the addition of pentoxifylline to a steroid regimen is effective in treating deteriorating muscle strength by comparing the muscle strength of PTX treated subjects and placebo treated subjects.

DETAILED DESCRIPTION:
DMD is the most common and devastating type of muscular dystrophy (incidence 1 in 3500 live born males worldwide). DMD is characterized by a complete loss of dystrophin, leading to progressive muscle weakness and wasting.

No cure is currently available despite our present understanding of the disorder and the discovery and characterization of the causative gene and its protein product dystrophin in 1987. Corticosteroids (prednisone, deflazacort) may delay disease progression and until now it is the only treatment that proved to be beneficial for patients with DMD. Other alternative supplements like creatine and glutamine also delay diseased progression.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 7 years to 100 years
* Ability to ambulate for 10 meters. Assistive devices are allowed.
* Diagnosis of DMD confirmed by at least one the following:
* On stable dose of prednisone, prednisolone or deflazacort for at least 12 months prior to screening.
* Participants who are on stable dose of any combination of the following compounds (creatine, glutamine, coenzyme Q10, vitamin E, C or D, JUVEN, arginine, calcium) must have taken these medications for at least 2 months prior to screening. Subjects are not required to take these medications to participate in the study.
* All other herbs, supplements or green tea (other than those noted above) have been discontinued 3 months prior to screening.
* Ability to provide reproducible QMT bicep score with no more than 15% variation between scores during screening.
* Normal blood clotting ability evidenced by a platelet function assessment (PFA).

Exclusion Criteria:

* Currently enrolled in another treatment clinical trial.
* History of significant concomitant illness or significant impairment of renal or hepatic function.
* History of impairment of blood clotting ability (as evidenced by increased PT/PTT or PFA over the upper limit of normal (ULN)).
* Recent cerebral or retinal hemorrhage.
* History of bleeding diathesis or gastric ulcer.

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Quantitative muscle strength will be measured using a CINRG Quantitative Muscle System (CQMS). The highest value of two consecutive maximal efforts will be recorded. The primary strength endpoint will be total CQMS score. | January 2008

SECONDARY OUTCOMES:
Strength of arm, leg and grip QMT scores Measured Screening and Months 1, 3, 6, 9 & 12 | January 2008
Manual Muscle Testing (MMT) score measured at screening and months 1, 3, 6, 9 & 12 using the Medical Research Council (MRC) scoring system. | January 2008
Functional evaluations measured at screening and months 1, 3, 6, 9 & 12 | January 2008
Time function assessments, including time rising from the floor, time to climb four standard stairs, and time to walk 10 meters. They will be measured at screening and months 1, 3, 6, 9 & 12. | January 2008
pulmonary function test (PFA's) measured at screening and months 1, 3, 6, 9 & 12 | January 2008
Pediatric Quality of Life (PQOL) measured at screening and months 1, 3, 6, 9 & 12 | January 2008
Goniometry measured at screening and months 1, 3, 6, 9 & 12 | January 2008
TNF-alpha and TGF-beta measured at screening and months 1, 3, 6, 9 & 12 | February 2008

CONTACTS AND LOCATIONS:
Overall Officials: Diana Escolar, MD, Study Chair — Children's National Medical Center, Center for Genetic Medicine
Locations (11):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
- Hospital Frances, Buenos Aires, Argentina
- Children's Hospital, Melbourne, Victoria, Australia
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
- Hadassah Hospital, Mt. Scopus, Jerusalem, Israel
- IRCCS C Mondino Foundation, Pavia, Italy, Italy

REFERENCES:
- See also: Related Info — http://www.cinrgresearch.org